CLINICAL TRIAL: NCT01263652
Title: The Relationship Between Patient Preferences, Analgesic Delivery Method and Pain Reduction in Spine Patients
Brief Title: Patient Preferences, Analgesic Delivery Method and Pain Reduction in Spine Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: inability to complete recruitment as planned
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Nimrod Rahamimov, Investigator, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SpinePainIMPO
Record Dates: First submitted 2010-10-06; First posted 2010-12-21 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Pain Relief
Keywords: Pain; intramuscular; oral; spine; preference
MeSH Terms: conditions — Pain | interventions — diclofenac hydroxyethylpyrrolidine; Diclofenac; Orphenadrine; Indomethacin; Tramadol; Dipyrone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMmed (Active Comparator): Patients receiving intra-muscular medication and oral placebo
  Interventions: Drug: Diclofenac hydroxyethylpyrrolidine; Drug: orphenadrine; Drug: Tramadol; Drug: Dipyrone
- POmed (Active Comparator): Patients receiving intra-muscular placebo and oral medication
  Interventions: Drug: Diclofenac hydroxyethylpyrrolidine; Drug: orphenadrine; Drug: Tramadol; Drug: Dipyrone

INTERVENTIONS:
Drug: Diclofenac hydroxyethylpyrrolidine — IM/PO
  Other Names: Voltaren, Abitren
Drug: orphenadrine — IM/PO orphenadrine
  Other Names: Flexin
Drug: Tramadol — IM/PO tramadol
  Other Names: Tramadex, Tramal
Drug: Dipyrone — PO/IM Dipyrone
  Other Names: Optalgin, Phanalgin

SUMMARY:
The investigators will conduct a randomized double blind study, to determine whether patient analgesic delivery mode preference affects pain reduction quality in non-surgical spine patients.

The patients will receive both intra-muscular and oral non-narcotic analgesics and placebo. During the study period, pain reduction parameters will be collected. At the end of the study period, the investigators will attempt to find a correlation between pre-study patient preferences and the quality of the pain reduction achieved.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic and acute back pain

Exclusion Criteria:

* Recent Spine Surgery

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12-31 (Estimated); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
pain scores on visual analog scale | visual analog scale will be mesuered before and one hour following every pain medication delivery
  up to 7 days for each patient per hospitalization

SECONDARY OUTCOMES:
Patient Questionnaire assessing pain and pain relief | Before administaration of pain control medication and one hour following analgesic administration
  A questionnaire will be filled immediately before and one hour following analgesic administration
patient preference Questionnaire | before first analgesic administration at the current hositalization
  every patient will be asked for his prefered analgesic delivery method

CONTACTS AND LOCATIONS:
Overall Officials: Nimrod Rahamimov, M.D., Principal Investigator — Western Galilee Hospital